CLINICAL TRIAL: NCT00186381
Title: Autologous Bone Marrow Transplantation for Acute Non-Lymphoblastic Leukemia During First or Subsequent Remission
Brief Title: Autologous Bone Marrow Transplantation in Acute Non-Lymphoblastic Leukemia During First or Subsequent Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Laura Johnston, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT8N; 77045; BMT8N; NCT00186381
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Leukemia, Myelocytic, Acute; Leukemia; Blood and Marrow Transplant (BMT)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

INTERVENTIONS:
Procedure: high dose chemotherapy then autologous hematopoietic cell transplant

SUMMARY:
Evaluate the role of high dose chemotherapy with autologous hematopoietic cell transplantation for AML.

DETAILED DESCRIPTION:
To use high dose chemotherapy with autologous stem cell rescue to try to increase the chance of long term control and cure of the disease.

ELIGIBILITY:
Inclusion Criteria:- must be in remission

* adequate organ function Exclusion Criteria:- prior MDS
* active infection
* liver disease

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1995-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Disease free survival (DFS)

SECONDARY OUTCOMES:
Transplant related mortality (TRM)
Toxicity
Adequacy of cell collections
Engraftment kinetics

CONTACTS AND LOCATIONS:
Overall Officials: Laura Johnston, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States